CLINICAL TRIAL: NCT01299805
Title: A Phase 1, Single-Center, Randomized, Single-Blind, Placebo-Controlled, Multiple-Dose Study to Assess the Effects of Oral Administration of Lu AA21004 20 mg on the Concentrations of Selected Neurotransmitters in Healthy Male Subjects
Brief Title: Effects of Vortioxetine (Lu AA21004) on the Concentrations of Selected Neurotransmitters in Healthy Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: LuAA21004_124; U1111-1119-1680 (Registry Identifier: WHO)
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Drug Therapy; pharmacodynamic
MeSH Terms: interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vortioxetine (Experimental): Vortioxetine 20 mg, encapsulated tablet, orally, once daily for up to 14 days.
  Interventions: Drug: Vortioxetine
- Placebo (Placebo Comparator): Vortioxetine placebo-matching capsules, orally, once daily for up to 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine — Encapsulated tablet
  Other Names: Lu AA21004; Brintellix
  Arms: Vortioxetine
Drug: Placebo — Vortioxetine placebo-matching capsules.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamics (the drug's effect on the body), the pharmacokinetics (the body's handling of the drug), and the safety and tolerability of vortioxetine, once daily (QD) in healthy men.

DETAILED DESCRIPTION:
This study will look at an investigational medicine called vortioxetine to see how the drug affects the body and how the body handles the drug.

The study enrolled 17 patients. Participants were randomly assigned at a 2:1 ratio to one of the following two treatment groups-which remained undisclosed to both the participant and study doctor during the study (unless there was an urgent medical need):

* Vortioxetine 20 mg
* Placebo (dummy inactive pill) - this was a capsule that looked like the study drug but had no active ingredient.

All participants were asked to take one capsule at the same time each day throughout the study.

This single-center trial was conducted in the United States. The overall time to participate in this study was approximately 7 weeks. Participants made 2 visits to the clinic, including 18 days confinement to the clinic, and were contacted by telephone 1 day and 27 days after leaving confinement for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Weighs at least 50 kg and has a body mass index between 19.0 and 32.0 kg/m^2, inclusive at Screening.
* Males who are nonsterilized and sexually active with a female partner of childbearing potential must agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 6 weeks after last dose of study medication. The acceptable method of contraception is defined as one that has no higher than a 1% failure rate.

Exclusion Criteria:

* Received any investigational compound within 45 days prior to Check-in (Day -2).
* Received Lu AA21004 in previous clinical study or as therapeutic agent.
* History of or uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, central nervous system, hepatic hematopoietic disease, renal metabolic, gastrointestinal, or endocrine disease, serious allergy, asthma, hypoxemia, hypertension, seizures, allergic skin rash or other abnormality, which may impact the ability of the participant to participate or potentially confound study results.
* Participant has 1 or more of the following:

  * Any current psychiatric disorder as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision (DSM-IV-TR).
  * Current or history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
  * Presence or history of a clinically significant neurological disorder (including epilepsy).
  * Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).
  * Any Axis II disorder.
* Has a known hypersensitivity to any component of the formulation of Lu AA21004.
* Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -2).
* Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular consumption of 4 or more units per day) within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. One unit is equivalent to a half-pint of beer or 1 measure of spirits or 1 glass of wine.
* The participant intends to impregnate or donate sperm during the course of this study or for 6 weeks after last dose.
* Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (e.g., a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis; frequent (more than once per week) occurrence of heartburn, or any intra-abdominal surgery (except laparoscopic cholecystectomy or uncomplicated appendectomy).
* Has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin that has not been in remission for at least 5 years prior to Day 1.
* Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody at Screening or a known history of human immunodeficiency virus infection.
* Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in (Day -2) or is unwilling to abstain from these products for the duration of the study.
* Cotinine test is positive at Screening or Check-in (Day 2).
* Has poor peripheral venous access.
* Has donated or lost 450 mL or more of his blood volume (including plasmapheresis), or had a transfusion of any blood product within 30 days prior to Day 1.
* Has a Screening or Check-in (Day -2) abnormal (clinically significant) electrocardiogram (ECG). Entry of any patient with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator.
* Has abnormal Screening or Day -2 laboratory values that suggest a clinically significant underlying disease or with the following lab abnormalities: alanine aminotransferase and/or aspartate aminotransferase >1.5 times the upper limit of normal.
* Has had cerebrospinal fluid (CSF) collection performed within 30 days prior to Check-in (Day -2).
* Has taken any selective serotonin reuptake inhibitor (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), or monoamine oxidase inhibitors, antipsychotics, tricyclic antidepressants, or mood stabilizers within the last year prior to Screening.
* Has a known hypersensitivity to the anesthetic or its derivatives used during CSF collection, or any medication used to prepare the area of lumbar puncture.
* Has significant vertebral deformities (scoliosis or kyphosis) which, in the opinion of the investigator, may interfere with lumbar puncture procedure.
* Has a history of clinically significant back pain and/or injury.
* Has local infection at the puncture site.
* Has a history of significant bleeding or coagulation disorder and/or low platelet levels (<130x10^9/L) or increased international normalized ratio (INR) (>1.3) at Screening.
* Answers positive to any suicidal ideation and/or suicidal behavior questions during administration of the Columbia-Suicide Severity Rating Scale.
* Has an orthostatic blood pressure drop of ≥20 mm Hg (based on the drop between supine and standing [3 minutes] systolic blood pressure) at Screening or Check-in (Day -2).
* Has abnormal Screening or Day -2 vital signs: resting systolic blood pressure ≤90 or ≥140 mm Hg or a resting diastolic blood pressure ≤50 or ≥90 mm Hg in supine position; resting pulse or heart rate (as read on ECG) <45 bpm or >100 bpm. No more than 2 repeat measurements.
* Exercises extensively in his normal life (e.g., marathon running, triathlon, physical sports at a contest level etc).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (1):
- Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in the United States from 14 March 2011 to 11 June 2011.
Pre-assignment Details: In this study, 17 healthy men were enrolled and randomized to receive an oral dose of vortioxetine 20 mg or placebo in a 2:1 ratio.
Period: Overall Study
Arm/Group | Vortioxetine | Placebo
Started | 12 | 5
Completed | 10 | 5
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vortioxetine | Placebo | Total
Number analyzed (Participants) | 12 | 5 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 34.3 (11.19) | 34.8 (10.71) | 34.4 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 5 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 9 | 5 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3 | 1 | 4
  White | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 5 | 17
Height [Mean (Standard Deviation); unit: cm] | 176.8 (5.88) | 175.9 (8.15) | 176.6 (6.37)
Weight [Mean (Standard Deviation); unit: kg] | 81.8 (8.84) | 79.9 (7.52) | 81.3 (8.29)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (2.85) | 25.8 (1.92) | 26.1 (2.56)
Current nicotine user [Number; unit: participants]
  Yes | 0 | 0 | 0
  No | 12 | 5 | 17
Former nicotine user [Number; unit: participants]
  Yes | 1 | 1 | 2
  No | 11 | 4 | 15
Drinking habits [Number; unit: participants]
  Drinks 0-14/week | 12 | 5 | 17
  Drinks >14/week | 0 | 0 | 0
Caffeine consumption [Number; unit: participants]
  Consumes 0-5 cups daily | 12 | 5 | 17
  Consumes >5 cups daily | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Effect Curve From Time Zero to 24 Hours Postdose of 5-hydroxytryptamine (5-HT) in Plasma
Description: The area under the effect-time curve from time 0 to 24 hours postdose (AUEC[0-24]) of the neurotransmitter 5-HT (serotonin) in plasma was measured at Baseline, after a single dose (Day 1) and after multiple doses (Day 14).
Time Frame: Day -1 (Baseline), Day 1 and Day 14. Blood samples were taken predose (up to 15 minutes prior) and at 1, 2, 4, 8, 12, 16 and 24 hours post-dose.
Population: The pharmacodynamic (PD) set consisted of all participants in the safety set with sufficient plasma or serum or CSF data for derivation of at least 1 PD parameter. If a patient's concentration profile contained ≤3 data points, the PD parameter results were not included. "n" indicates the number of patients with available data at each time point.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
pg*hr/mL
  Day -1 (n=10, 4) | 4183024 (1362135) | 3854399 (1728230)
  Day 1 (n=6, 4) | 4224058 (2028835) | 3912292 (2083773)
  Day 14 (n=9, 5) | 1718863 (530633) | 3858350 (2212719)

2. Primary Outcome: Maximum Concentration of 5-HT in Plasma
Description: The maximum observed effect (Emax), assessed by the maximum observed concentration of 5-HT in plasma measured at Baseline, after a single dose (Day 1) and after multiple doses (Day 14).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
pg/mL
  Day -1 (n=10, 4) | 273800 (111197) | 231500 (98083.3)
  Day 1 (n=6, 4) | 247667 (136695) | 251250 (63615.4)
  Day 14 (n=9, 5) | 94233.3 (40258.4) | 242200 (115103)

3. Primary Outcome: Time to Maximum Concentration of 5-HT in Plasma
Description: The time to reach maximum pharmacodynamic effect (Emax) was assessed by the time to maximum concentration of 5-HT in plasma at Baseline, after a single dose (Day 1) and after multiple doses (Day 14).
Time Frame: Day -1 (Baseline), Day 1 and Day 14. Blood samples were taken predose and at 1, 2, 4, 8, 12, 16, and 24 hours postdose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
hours
  Day -1 (n=10, 4) | 12.65 (9.409) | 7.26 (7.984)
  Day 1 (n=6, 4) | 4.86 (7.253) | 14.42 (11.146)
  Day 14 (n=9, 5) | 9.11 (10.080) | 8.40 (6.986)

4. Primary Outcome: Area Under the Effect Curve From Time Zero to 24 Hours Postdose of 5-HT in Cerebrospinal Fluid
Description: The area under the effect-time curve from time 0 to 24 hours postdose (AUEC[0-24]) of 5-hydroxytryptamine (5-HT) in cerebrospinal fluid (CSF) was measured at Baseline, after a single dose (Day 1) and after multiple doses (Day 14).
Time Frame: Day -1 (Baseline), Day 1 and Day 14. CSF samples were taken prior to dose and at 1, 2, 4, 8, 12, 16, and 24 hours postdose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
pg*hr/mL
  Day -1 (n=11, 5) | 987.71 (1898.943) | 509.77 (199.658)
  Day 1 (n=11, 5) | 627.78 (164.679) | 497.40 (302.720)
  Day 14 (n=9, 5) | 1165.73 (290.389) | 444.88 (24.908)

5. Primary Outcome: Maximum Concentration of 5-HT in Cerobrospinal Fluid
Description: The maximum observed effect (Emax), assessed by the maximum concentration of 5-HT in cerebrospinal fluid (CSF) measured at Baseline, after a single dose (Day 1) and after multiple doses (Day 14).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
pg/mL
  Day -1 (n=11, 5) | 116.60 (293.721) | 67.74 (94.396)
  Day 1 (n=11, 5) | 35.46 (13.172) | 24.10 (14.030)
  Day 14 (n=9, 5) | 59.80 (16.524) | 51.46 (33.647)

6. Primary Outcome: Time to Maximum Concentration of 5-HT in Cerebrospinal Fluid
Description: The time to reach maximum pharmacodynamic effect (Emax) was assessed by the time to maximum concentration of 5-HT in cerebrospinal fluid (CSF) at Baseline, after a single dose (Day 1) and after multiple doses (Day 14).
Time Frame: Day -1, Day 1 and Day 14. CSF samples were taken predose and at 1, 2, 4, 8, 12, 16, and 24 hours postdose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
hours
  Day -1 (n=11, 5) | 4.30 (5.890) | 7.13 (10.624)
  Day 1 (n=11, 5) | 17.32 (7.177) | 6.92 (8.225)
  Day 14 (n=9, 5) | 3.02 (3.576) | 4.94 (6.964)

7. Primary Outcome: Area Under the Effect Curve From Time Zero to 24 Hours Postdose of 5-hydroxyindoleacetic Acid (5-HIAA) in Plasma
Description: Area under the effect-time curve from time 0 to 24 hours postdose (AUEC[0-24]) of 5-HIAA, a metabolite of the neurotransmitter serotonin, in plasma was measured after a single dose (Day 1) and after multiple doses (Day 14). Note: Plasma samples for 5-HIAA on Day -1 were lost in shipping. Therefore, no PD parameters were calculated for Day -1.
Time Frame: Day 1 and Day 14. Blood samples were taken predose and at 1, 2, 4, 8, 12, 16 and 24 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
ng*hr/mL
  Day 1 (n=12, 5) | 140.01 (23.633) | 145.92 (28.844)
  Day 14 (n=10, 5) | 143.69 (30.049) | 140.40 (25.305)

8. Primary Outcome: Maximum Concentration of 5-HIAA in Plasma
Description: The maximum observed effect (Emax), assessed by the maximum observed concentration of 5-HIAA in plasma measured after a single dose (Day 1) and after multiple doses (Day 14). Note: Plasma samples for 5-HIAA on Day -1 were lost in shipping. Therefore, no PD parameters were calculated for Day -1
Time Frame: Day 1 and Day 14. Blood samples were taken predose (up to 15 minutes prior) and at 1, 2, 4, 8, 12, 16 and 24 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
ng/mL
  Day 1 (n=12, 5) | 7.25 (1.113) | 6.97 (1.282)
  Day 14 (n=10, 5) | 6.90 (1.402) | 7.10 (1.301)

9. Primary Outcome: Time to Maximum Concentration of 5-HIAA in Plasma
Description: The time to reach maximum pharmacodynamic effect (Emax) was assessed by the time to maximum concentration of 5-hydroxyindoleacetic acid (5-HIAA) in plasma after a single dose (Day 1) and after multiple doses (Day 14). Note: Plasma samples for 5-HIAA on Day -1 were lost in shipping. Therefore, no PD parameters were calculated for Day -1.
Time Frame: Day 1 and Day 14. Blood samples were taken predose and at 1, 2, 4, 8, 12, 16 and 24 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
hours
  Day 1 (n=12, 5) | 13.02 (10.992) | 15.13 (9.886)
  Day 14 (n=10, 5) | 16.80 (7.005) | 18.40 (5.367)

10. Primary Outcome: Area Under the Effect Curve From Time Zero to 24 Hours Postdose of 5-HIAA in Cerebrospinal Fluid
Description: The area under the effect-time curve from time 0 to 24 hours postdose (AUEC[0-24]) of 5-hydroxyindoleacetic acid (5-HIAA) in cerebrospinal fluid (CSF) was measured at Baseline, after a single dose (Day 1) and after multiple doses (Day 14).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
ng*hr/mL
  Day -1 (n=12, 5) | 620.61 (182.391) | 718.14 (247.082)
  Day 1 (n=12, 5) | 636.14 (246.071) | 774.95 (319.860)
  Day 14 (n=9, 5) | 429.23 (99.575) | 644.24 (206.121)

11. Primary Outcome: Maximum Concentration of 5-HIAA in Cerebrospinal Fluid
Description: The maximum observed effect (Emax), assessed by the maximum observed concentration of 5-HIAA in cerebrospinal fluid (CSF) measured at Baseline, after a single dose (Day 1) and after multiple doses (Day 14).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
ng/mL
  Day -1 (n=12, 5) | 29.87 (8.231) | 34.30 (12.270)
  Day 1 (n=12, 5) | 31.13 (9.567) | 36.98 (18.346)
  Day 14 (n=9, 5) | 20.18 (4.935) | 30.16 (8.768)

12. Primary Outcome: Time to Maximum Concentration of 5-HIAA in Cerebrospinal Fluid
Description: The time to reach maximum pharmacodynamic effect (Emax) was assessed by the time to maximum concentration of 5-hydroxyindoleacetic acid (5-HIAA) in cerebrospinal fluid (CSF) at Baseline, after a single dose (Day 1) and after multiple doses (Day 14).
Time Frame: Day -1, Day 1 and Day 14. CSF samples were taken prior to dose and at 1, 2, 4, 8, 12, 16, and 24 hours postdose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 12 | 5
hours
  Day -1 (n=12, 5) | 14.16 (10.710) | 19.78 (8.877)
  Day 1 (n=12, 5) | 6.24 (8.960) | 19.00 (10.621)
  Day 14 (n=9, 5) | 11.70 (10.576) | 9.90 (9.592)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vortioxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/5
Other Adverse Events (participants affected / at risk) | 11/12 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=12) | Placebo (N=5)
Nausea (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Chest discomfort (General disorders) | 1 | 0
Tenderness (General disorders) | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights therefrom or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.